CLINICAL TRIAL: NCT01940718
Title: Androgen Regulation of Priapism in Sickle Cell Disease
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Funding could not be secured
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00076088
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Priapism; Sickle Cell Disease; Hypogonadism
Keywords: Priapism; Sickle cell disease; Testosterone; Androgen deficiency
MeSH Terms: conditions — Priapism; Anemia, Sickle Cell; Hypogonadism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transdermal Testosterone (Experimental): Transdermal Androgel 1.62% (20.25 mg testosterone = 1 pump actuations) to be applied once daily for 3.5 months. Initial dose will be at lowest level, 20.25 mg testosterone with dosing adjustments given in 20.25 mg testosterone increments.
  Interventions: Drug: Transdermal Androgel

INTERVENTIONS:
Drug: Transdermal Androgel — T dosing will be initiated at the lowest possible level (20.25 mg testosterone = 1 pump actuation) which is expected to increase average serum T concentrations no higher than the mid-normal range (500-800 ng/dl), with respect to expected baseline measurements in our population (~300-500 ng/dl).The T dose will be adjusted two weeks after initiation of treatment based on the measurement of serum T levels. Dosing adjustments can be made at 20.25 mg testosterone increments. The medication will be taken transdermally once daily for 3.5 months.
  Other Names: Androgel 1.62%

SUMMARY:
It is believed that when androgen (testosterone) levels are below normal there is a disturbance of normal bodily functioning that is associated with priapism in some men. Conversely, it is believed that testosterone replacement will improve the condition of priapism when the testosterone levels are brought to normal. In turn, this will also improve psychological well being in men with sickle cell disease (SCD).

DETAILED DESCRIPTION:
The central hypothesis of this proposal is that a decline in androgen levels results in decreased action and contributes to the molecular derangements associated with priapism. Optimizing androgen status may promote regulatory molecular mechanisms that protect against priapism. This clinical trial will investigate the potential benefit of precise testosterone replacement for ameliorating priapism and improving psychological well-being in hypogonadal men with SCD.

This clinical trial aims to evaluate the efficacy of testosterone replacement therapy on the frequency of recurrent priapism in patients with SCD. The sub-hypothesis that testosterone (T) replacement to achieve serum T concentrations at a target range reduces recurrent priapism will be tested. This aim will involve subjective and objective assessments of priapism occurrences and erectile ability including priapism inventory instruments, standardized questionnaires of erectile function (EF) and quality of life, and Rigiscan™ erection monitoring in a 3.5-month pilot investigation.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-50
* History of SCD
* Episodes of prolonged penile erection in the absence of sexual interest or desire, with an average frequency of at least twice weekly, when averaged over the previous four weeks
* serum testosterone level below 550 ng/dl
* Ability to provide informed consent

Exclusion Criteria:

* Alcohol use exceeding two standard drinks daily
* Prostate conditions including prostate specific antigen (PSA) elevation (>2.5 ng/ml)
* Known sleep apnea
* Known cirrhosis
* Enlarged and painful male breasts

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
change in frequency of priapism episodes | Baseline to 3 months post intervention
  A "Priapism sexual activity log" will be administered to participants. In the log, participants will be asked to quantify the number of priapic episodes they have experienced in the previous 2 weeks according to the following scale/tiers: 0 = no episodes, 1 = 1-2 episodes, 2 = 3-4 episodes, 3 = 5-8 episodes and 6 = greater than 20 episodes.

SECONDARY OUTCOMES:
change in quality of life | Baseline to 3 months post intervention
  The RAND 12 questionnaire will be administered. This is a validated questionnaire evaluating the patient's perception of their overall health.
change in quality of erections | Baseline to 3 months post intervention
  The RigiScan will be used. This is an external instrument to measure penile tumescence and rigidity
change in EF | Baseline to 3 months post intervention
  The International Index of Erectile Function (IIEF) will be administered. This is a 15 item questionnaire . The questionnaire measures Erectile Function (scored from 0-30), Intercourse satisfaction (0-15), orgasmic function (0-10), Sexual Desire (2-10) and Overall satisfaction (2-10).

CONTACTS AND LOCATIONS:
Overall Officials: Arthur L Burnett, MD, MBA, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Johns Hopkins Hospital, Baltimore, Maryland, United States